CLINICAL TRIAL: NCT04516720
Title: Creation of a Clinical Database on Primary Nervous System Tumors
Acronym: BDD-NO
Status: Recruiting | Type: Observational
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Other Study IDs: PROICM 2017-01 BNO
Record Dates: First submitted 2020-08-11; First posted 2020-08-18 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Nervous System Tumor
Keywords: Primary central nervous system tumors; clinical database
MeSH Terms: conditions — Nervous System Neoplasms | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary Nervous System Tumors arm: The information letter will be delivered by the investigator physician to the patients to inform them on the study, its implementation and their complete freedom to participate or not.
  Clinical Data and Questionnaires:
  1. For the retrospective part
     * Patient identification based on data from the Medical Information Department (DIM) of the ICM;
     * Verification of the eligibility criteria;
     * Inclusion of patients in a coded form in BDD-NO;
     * Implementation of the database with the data already collected (as an coded EXCEL file) in specific studies (some patients are included in several of these studies): study of diffuse low grade gliomas, study on anaplastic gliomas, study on the place of Bevacizumab in high-grade gliomas, clinical database created
     * Collection of clinical data from each patient's medical record
  2. For the prospective part
     * Inclusion of patients in a coded form in BDD-NO;
     * Collection of clinical data from each patient's medical record.
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — Diagnostic data : date and description of first symptoms,date of radiological diagnosis, tumor localization, number of lesions, date of histological diagnosis, histological diagnostic mode, histological diagnosis, WHO grade (I, II, III or IV), immunohistochemic data, molecular alterations therapeutic sequence : type of treatment, baseline exam before each treatment, surgery, radiothérapy, systemic treatment, clinical study, follow up until death

SUMMARY:
the creation of a clinical database including data for all PCNST patients is of high interest. This database will allow us to develop clinical studies on:

* The clinical, radiological and biological presentation of tumors, the impact of oncological treatments and the evaluation of survival for the different subtypes of Primary central nervous system tumors (PCNST). This is particularly important for rare histological subtypes of PCNST for which the current knowledge is scarce;
* Clinical, radiological and biological factors predictive of tumor response to treatments;
* Prognostic factors.

DETAILED DESCRIPTION:
Primary central nervous system tumors (PCNST) correspond to all primitive tumors involving central nervous system structures, meninges and the origin of the cranial and paraspinal nerves. They have a malignant, benign, or borderline evolution. TPSNC represent a heterogeneous group of tumors, with more than 140 subtypes described in the WHO classification. The causes, prognostic factors, and therapeutic management differ according to the histological subtype.

The incidence of all of TPSNCs ranges from 17.6 to 22.0/105 in North American and European studies. However, because of the high number of different histological subtypes, most of them must be considered as rare tumors. Moreover, they represent a major public health problem due to high morbidity [8] and mortality.

In this context, the creation of a clinical database including data for all PCNST patients is of high interest. This database will allow us to develop clinical studies on:

* The clinical, radiological and biological presentation of tumors, the impact of oncological treatments and the evaluation of survival for the different subtypes of PCNST. This is particularly important for rare histological subtypes of PCNST for which the current knowledge is scarce;
* Clinical, radiological and biological factors predictive of tumor response to treatments;
* Prognostic factors.

The database will also allow us to develop or participate in multicentric clinical studies, at the national or international level, as well as to facilitate the identification of patients for inclusion in translational studies

ELIGIBILITY:
Inclusion Criteria:

* Adult patient aged ≥ 18, no age limit;
* Diagnosis of Primary central nervous system tumors ;
* Patient treated at the Montpellier Cancer Institute, whatever the treatment received (systemic treatment, radiotherapy or exclusive supportive care);
* For the retrospective part of the study, patient first treated at the Montpellier Cancer Institute between January 1rst, 2004 and the beginning of the prospective part;
* Patient information for the retrospective (patient still alive at the beginning of the study) and prospective study.

Exclusion Criteria:

* Secondary lesions of the central nervous system;
* Patient not affiliated to a social protection scheme;
* Subject under tutelage, curatorship or safeguard of justice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patient with Primary central nervous system tumors and treated at the Montpellier Cancer Institute
Sampling Method: Probability Sample
Enrollment: 1700 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2035-01 (Estimated); Study Completion 2039-01 (Estimated)

PRIMARY OUTCOMES:
Establish an exhaustive database of patients treated for a Primary central nervous system tumors at the Montpellier Cancer Institute, whatever the histological subtype and the oncological treatment | From date of inclusion until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  collection of clinical data in the medical record

SECONDARY OUTCOMES:
Realization of clinical studies specific to certain histological subtypes to be carried out on the clinical, radiological and biological presentation of patients, specific oncological treatments and toxicities, prognostic factors and survival data | From date of inclusion until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  obtaining reliable clinical data for write new clinical trials project
To allow the realization of epidemiological studies specific to certain histological subtypes | From date of inclusion until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  new clinical trials project based on this clinical database
To facilitate the identification of patients for inclusion in French or European retrospective studies | From date of inclusion until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  new clinical trials project based on this clinical database

CONTACTS AND LOCATIONS:
Overall Officials: Amélie DARLIX, MD, Study Chair — Institut régional du Cancer Montpellier
Locations (1):
- Icm Val D'Aurelle, Montpellier, Herault, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Louis DN, Ohgaki H, Wiestler OD, Cavenee WK, Burger PC, Jouvet A, Scheithauer BW, Kleihues P. The 2007 WHO classification of tumours of the central nervous system. Acta Neuropathol. 2007 Aug;114(2):97-109. doi: 10.1007/s00401-007-0243-4. Epub 2007 Jul 6. PMID 17618441
- [Result] Louis DN, Perry A, Reifenberger G, von Deimling A, Figarella-Branger D, Cavenee WK, Ohgaki H, Wiestler OD, Kleihues P, Ellison DW. The 2016 World Health Organization Classification of Tumors of the Central Nervous System: a summary. Acta Neuropathol. 2016 Jun;131(6):803-20. doi: 10.1007/s00401-016-1545-1. Epub 2016 May 9. PMID 27157931
- [Result] Ostrom QT, Gittleman H, Fulop J, Liu M, Blanda R, Kromer C, Wolinsky Y, Kruchko C, Barnholtz-Sloan JS. CBTRUS Statistical Report: Primary Brain and Central Nervous System Tumors Diagnosed in the United States in 2008-2012. Neuro Oncol. 2015 Oct;17 Suppl 4(Suppl 4):iv1-iv62. doi: 10.1093/neuonc/nov189. Epub 2015 Oct 27. No abstract available. PMID 26511214
- [Result] Wohrer A, Waldhor T, Heinzl H, Hackl M, Feichtinger J, Gruber-Mosenbacher U, Kiefer A, Maier H, Motz R, Reiner-Concin A, Richling B, Idriceanu C, Scarpatetti M, Sedivy R, Bankl HC, Stiglbauer W, Preusser M, Rossler K, Hainfellner JA. The Austrian Brain Tumour Registry: a cooperative way to establish a population-based brain tumour registry. J Neurooncol. 2009 Dec;95(3):401-411. doi: 10.1007/s11060-009-9938-9. Epub 2009 Jun 28. PMID 19562257
- [Result] Baldi I, Gruber A, Alioum A, Berteaud E, Lebailly P, Huchet A, Tourdias T, Kantor G, Maire JP, Vital A, Loiseau H; Gironde TSNC Registry Group. Descriptive epidemiology of CNS tumors in France: results from the Gironde Registry for the period 2000-2007. Neuro Oncol. 2011 Dec;13(12):1370-8. doi: 10.1093/neuonc/nor120. Epub 2011 Oct 6. PMID 21980160
- [Result] Crocetti E, Trama A, Stiller C, Caldarella A, Soffietti R, Jaal J, Weber DC, Ricardi U, Slowinski J, Brandes A; RARECARE working group. Epidemiology of glial and non-glial brain tumours in Europe. Eur J Cancer. 2012 Jul;48(10):1532-42. doi: 10.1016/j.ejca.2011.12.013. Epub 2012 Jan 7. PMID 22227039
- [Result] Darlix A, Zouaoui S, Rigau V, Bessaoud F, Figarella-Branger D, Mathieu-Daude H, Tretarre B, Bauchet F, Duffau H, Taillandier L, Bauchet L. Epidemiology for primary brain tumors: a nationwide population-based study. J Neurooncol. 2017 Feb;131(3):525-546. doi: 10.1007/s11060-016-2318-3. Epub 2016 Nov 16. PMID 27853959
- [Result] DeAngelis LM. Brain tumors. N Engl J Med. 2001 Jan 11;344(2):114-23. doi: 10.1056/NEJM200101113440207. No abstract available. PMID 11150363
- [Result] Jakola AS, Skjulsvik AJ, Myrmel KS, Sjavik K, Unsgard G, Torp SH, Aaberg K, Berg T, Dai HY, Johnsen K, Kloster R, Solheim O. Surgical resection versus watchful waiting in low-grade gliomas. Ann Oncol. 2017 Aug 1;28(8):1942-1948. doi: 10.1093/annonc/mdx230. PMID 28475680
- [Result] Capelle L, Fontaine D, Mandonnet E, Taillandier L, Golmard JL, Bauchet L, Pallud J, Peruzzi P, Baron MH, Kujas M, Guyotat J, Guillevin R, Frenay M, Taillibert S, Colin P, Rigau V, Vandenbos F, Pinelli C, Duffau H; French Reseau d'Etude des Gliomes. Spontaneous and therapeutic prognostic factors in adult hemispheric World Health Organization Grade II gliomas: a series of 1097 cases: clinical article. J Neurosurg. 2013 Jun;118(6):1157-68. doi: 10.3171/2013.1.JNS121. Epub 2013 Mar 15. PMID 23495881
- [Result] Boetto J, Bertram L, Moulinie G, Herbet G, Moritz-Gasser S, Duffau H. Low Rate of Intraoperative Seizures During Awake Craniotomy in a Prospective Cohort with 374 Supratentorial Brain Lesions: Electrocorticography Is Not Mandatory. World Neurosurg. 2015 Dec;84(6):1838-44. doi: 10.1016/j.wneu.2015.07.075. Epub 2015 Aug 14. PMID 26283485
- [Result] Mandonnet E, Wager M, Almairac F, Baron MH, Blonski M, Freyschlag CF, Barone F, Fontaine D, Pallud J, Hegi M, Viegas C, Zetterling M, Spena G, Goodden J, Rutten GJ, Taillandier L, Foroglu N, Darlix A, Skrap M, Martino J, von Campe G, Madadaki C, Gayat E, de Witt Hamer P, Gil Robles S, Sarubbo S, Santarius T, Bello L, Forster MT, Duffau H. Survey on current practice within the European Low-Grade Glioma Network: where do we stand and what is the next step? Neurooncol Pract. 2017 Dec;4(4):241-247. doi: 10.1093/nop/npw031. Epub 2017 Jan 17. PMID 31386020